CLINICAL TRIAL: NCT07252544
Title: Isosorbide Mononitrate and Butylphthalide to Reduce the Risk of Disability in Patients With Acute Lacunar Stroke: a 2×2 Factorial Randomized Controlled Trial (IMPACT)
Brief Title: Isosorbide Mononitrate and Butylphthalide to Reduce the Risk of Disability in Patients With Acute Lacunar Stroke (IMPACT)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023ZD0504802
Record Dates: First submitted 2025-09-09; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Lacunar; Stroke, Acute Ischemic; Cerebral Small Vessel Diseases
MeSH Terms: conditions — Stroke, Lacunar; Ischemic Stroke; Cerebral Small Vessel Diseases | interventions — isosorbide-5-mononitrate; 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- isosorbide mononitrate plus butylphthalide (Experimental)
  Interventions: Drug: Isosorbide Mononitrate; Drug: Butylphthalide
- isosorbide mononitrate plus butylphthalide placebo (Experimental)
  Interventions: Drug: Isosorbide Mononitrate; Drug: Butylphthalide Placebo
- isosorbide mononitrate placebo plus butylphthalide (Experimental)
  Interventions: Drug: Butylphthalide; Drug: Isosorbide Mononitrate Placebo
- isosorbide mononitrate placebo plus butylphthalide placebo (Placebo Comparator)
  Interventions: Drug: Isosorbide Mononitrate Placebo; Drug: Butylphthalide Placebo

INTERVENTIONS:
Drug: Isosorbide Mononitrate — Days 1-7: Isosorbide mononitrate injection, 20 mg once daily by intravenous infusion.
  Days 8-6 months: Isosorbide mononitrate sustained-release tablets, 40 mg once daily orally (dose reduced to 20 mg once daily during the final week).
  Arms: isosorbide mononitrate plus butylphthalide; isosorbide mononitrate plus butylphthalide placebo
Drug: Butylphthalide — Days 1-7: Butylphthalide injection, 25 mg twice daily by intravenous infusion.
  Days 8-6 months: Butylphthalide soft capsules, 200 mg three times daily orally.
  Arms: isosorbide mononitrate placebo plus butylphthalide; isosorbide mononitrate plus butylphthalide
Drug: Isosorbide Mononitrate Placebo — Days 1-7: Isosorbide mononitrate injection placebo, once daily by intravenous infusion.
  Days 8-6 months: Isosorbide mononitrate sustained-release tablet placebo, once daily orally (dose reduced to half a tablet once daily during the final week).
  Arms: isosorbide mononitrate placebo plus butylphthalide; isosorbide mononitrate placebo plus butylphthalide placebo
Drug: Butylphthalide Placebo — Days 1-7: Butylphthalide injection placebo, twice daily by intravenous infusion.
  Days 8-6 months: Butylphthalide soft capsule placebo, 2 capsules three times daily orally.
  Arms: isosorbide mononitrate placebo plus butylphthalide placebo; isosorbide mononitrate plus butylphthalide placebo

SUMMARY:
The goal of this multicenter, double-blind, 2×2 factorial randomized controlled trial is to evaluate the efficacy and safety of isosorbide mononitrate, butylphthalide, and their combination in reducing disability in patients with acute lacunar stroke.

DETAILED DESCRIPTION:
There is an urgent need for effective therapeutic strategies for acute ischemic cerebral small vessel disease (CSVD). Isosorbide mononitrate and butylphthalide may exert protective effects; however, large-scale randomized controlled trials are required to confirm their efficacy and safety and to guide clinical practice.

In this study, patients presenting with a clinical lacunar syndrome within 7 days of onset will be randomly assigned, in a 1:1:1:1 ratio, to one of four groups in addition to routine care: (1) isosorbide mononitrate plus butylphthalide, (2) isosorbide mononitrate plus butylphthalide placebo, (3) isosorbide mononitrate placebo plus butylphthalide, or (4) isosorbide mononitrate placebo plus butylphthalide placebo. The treatment period will last 6 months, with a total follow-up of 1 year, including assessments at 7 days, 1 month, 3 months, 6 months, and 1 year.

The primary efficacy outcome is post-stroke disability at 6 months. The primary safety outcome is moderate or more severe headache within 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 30 years;
2. Clinical lacunar syndrome within 7 days;
3. Brain CT/MRI after symptom onset:

   1. a relevant (in time and location) acute lacunar infarct;
   2. if no relevant lesion, symptom duration >24 hours, with no other suspected stroke etiologies (such as cerebral hemorrhage, cortical infarction, seizures, etc.)
4. MoCA score meeting the following criteria:

   1. MoCA ≥ 13 if educated ≤ 6 years;
   2. MoCA ≥ 15 if 7 ≤ educated ≤ 12 years;
   3. MoCA ≥ 18 if educated ≥ 13 years；
5. mRS ≤ 1 prior to this episode;
6. Patient or a legally authorized representative signed informed consent.

Exclusion Criteria:

1. Ischemic stroke of large artery atherosclerosis, cardioembolism, or other etiologies (TOAST classification);
2. Diagnosed or suspected hereditary CSVD;
3. Intracerebral hemorrhage within the past 3 months including parenchymal, intraventricular, subarachnoid hemorrhage, subdural/epidural hematoma;
4. Neurodegenerative diseases or systemic diseases that may lead to cognitive impairment, such as Alzheimer's disease, mixed dementia, Parkinson's disease, systemic autoimmune diseases, hepatic encephalopathy, or uremic encephalopathy.
5. Previously diagnosed psychiatric disorders (DSM-5 criteria).
6. Other active neurological disorders (e.g., recurrent seizures, brain tumors, vascular malformations, untreated aneurysms >3 mm).
7. Hypotension (seated systolic blood pressure <100 mmHg), bradycardia (heart rate <60 bpm), sick sinus syndrome or severe cardiopulmonary disease.
8. History of congestive heart failure, acute myocardial infarction or other severe cardiac dysfunctions (NYHA Class III-IV).
9. Coagulation disorders, bleeding tendency or systemic bleeding, including but not limited to prothrombin time >3×upper limit of normal (ULN), platelet count <50×109/L, hemophilia, capillary fragility, gastrointestinal bleeding, urinary tract bleeding, hemoptysis, or vitreous hemorrhage, etc.
10. Severe hepatic or renal insufficiency (note: severe hepatic insufficiency is defined as ALT or AST > 3×ULN or acute hepatitis, chronic active hepatitis, cirrhosis; severe renal insufficiency is defined as eGFR < 45 ml/min/1.73m², creatinine clearance < 40 ml/min, or known chronic kidney disease of stage 3 or higher).
11. Head trauma, intracranial or spinal surgery, major surgical procedures or severe trauma within the past 4 weeks.
12. ISMN or NBP use within the past 3 days.
13. Have contraindications to ISMN or NBP, or allergy to their components.
14. Have to use the contraindicated drugs of this trial for a long time.
15. Pregnant, breastfeeding or planning to pregnant during this study.
16. Unable to tolerate MRI or with MRI contraindications.
17. Have severe diseases or expected survival <12 months.
18. Participate in other clinical trials within 30 days before this trial.
19. Unlikely to comply with study procedures and follow-up procedures for whatever reason in the opinion of the research physician.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3156 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with post-stroke disability at 6 months | 6 months
  A composite endpoint defined as the occurrence of any of the following: modified Rankin Scale (mRS) score ≥ 3, major adverse cardiovascular events (MACE), cognitive impairment, or all-cause mortality. The mRS measures post-stroke functional outcome on a scale from 0 (no symptoms) to 6 (death). MACE includes non-fatal stroke, non-fatal myocardial infarction (MI), and vascular death.The assessment of cognitive function involves three stages: a cognitive screening test, supplementary cognitive testing, and adjudication by an expert panel. The Beijing version of the Montreal Cognitive Assessment (MoCA) is used as the cognitive screening scale. Scores on the MoCA range from 0 to 30, with lower scores indicating greater cognitive impairment.The supplementary cognitive assessment includes the evaluation of several domains: executive function, attention and processing speed, language, and memory, as well as activities of daily living.
Incidence of moderate or more severe headache within 6 months | 6 months
  Headache severity is assessed using the Numerical Rating Scale (NRS), where: 0 indicates no pain; 1 represents a mild headache (including feelings of head pressure or throbbing that are not considered painful); a score of 4 or higher (≥4) represents a headache of at least moderate intensity; and 10 represents the worst headache imaginable to the subject.

SECONDARY OUTCOMES:
Proportion of participants with post-stroke disability at 1 year | 1 year
  The difinition of post-stroke disability is the same as the primary outcome measure.
Proportion of participants with the modified Rankin Scale (mRS) score ≥ 3 at 6 months and 1 year | 6 months and 1 year
  The modified Rankin Scale (mRS) is used to measure the degree of disability and dependence after a stroke. The scale ranges from 0 to 6. A score of 0 represents no symptoms, 1 represents no significant disability, 2 represents slight disability, 3 represents moderate disability, 4 represents moderately severe disability, 5 represents severe disability, and 6 represents death.
Incidence of recurrent stroke within 6 months and 1 year | 6 months and 1 year
Proportion of participants with dementia at 6 months and 1 year | 6 months and 1 year
  Dementia (all of the following criteria must be met):
  A. Evidence of significant cognitive decline from a previous level of performance in one or more cognitive domains (complex attention, executive function, learning and memory, language, perceptual-motor, or social cognition) based on:1.Concern from the individual, a knowledgeable informant, or the clinician that there has been a significant decline in cognitive function. 2.A substantial impairment in cognitive performance, preferably documented by standardized neuropsychological testing or, in its absence, another quantified clinical assessment.
  B. The cognitive deficits interfere with independence in everyday activities (i.e., at a minimum, requiring assistance with complex instrumental activities of daily living, such as paying bills or managing medications).
  C. The cognitive deficits do not occur exclusively in the context of a delirium.
  D. The cognitive deficits are not better explained by another mental disorder.
National Institutes of Health Stroke Scale (NIHSS) scores at 7 days, 6 months, and 1 year (including changes from baseline) | baseline, 7 days, 6 months, and 1 year
  The National Institutes of Health Stroke Scale (NIHSS) is a standardized tool used to objectively measure the severity of a stroke by quantifying a patient's neurological deficits. Its primary purposes are to evaluate the acuity of a stroke, guide treatment decisions, and predict patient outcomes. The scale's total score ranges from 0 to 42, with higher scores representing more severe neurological impairment.
Incidence of hypotension within 6 months | 6 months
  Hypotension is defined as a systolic blood pressure (SBP) of less than 100 mmHg or a 30% decrease from baseline.
Incidence of syncope within 6 months | 6 months
  Syncope is a transient loss of consciousness caused by transient global cerebral hypoperfusion, characterized by a rapid onset, short duration, and spontaneous, complete recovery.
  The diagnosis requires the following conditions to be met:
  1. A transient loss of consciousness with a rapid onset (from a few seconds to 1 minute);
  2. A short duration (from a few seconds to a few minutes);
  3. Spontaneous and complete recovery;
  4. Absence of focal neurological signs;
  5. Exclusion of head trauma and epileptic seizures.
Incidence of liver function impairment within 6 months | 6 months
  Liver function impairment may be diagnosed if at least one of the following criteria is met:
  1. Serum AST or ALT > 5 × the upper limit of normal (ULN), or ALP > 2 × ULN (or from an abnormal baseline value);
  2. Serum total bilirubin (TBil) > 2.5 mg/dL (42.75 μmol/L) accompanied by any elevation in serum AST, ALT, or ALP levels.
Incidence of any bleeding within 6 months | 6 months
  Bleeding events are evaluated using the GUSTO (Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries) classification and categorized as severe, moderate, or mild.
Incidence of symptomatic intracranial hemorrhage within 6 months | 6 months
  According to the Heidelberg Bleeding Classification established at the 12th Thrombolytic Therapy in Acute Ischemic Stroke workshop in Germany in 2015, symptomatic intracerebral hemorrhage (sICH) is defined as meeting all of the following conditions:
  1. Any form of intracranial hemorrhage (including types 1a, 1b, 1c, 2, 3a, 3b, 3c, and 3d of the Heidelberg classification) that is detected by imaging (head CT or MRI) and confirmed by a radiologist;
  2. The patient experiences clinical deterioration, defined as: an increase in the NIHSS score of ≥ 4 points from the last score prior to deterioration, OR an increase of ≥ 2 points on any single item of the NIHSS, OR an outcome leading to tracheal intubation, decompressive craniectomy, ventricular drainage, or other major medical/surgical intervention;
  3. The clinical deterioration cannot be explained by any cause other than the intracranial hemorrhage.

OTHER OUTCOMES:
≥ 80% of patients taking ≥ 50% of the trial dose up to 6 months | 6 months
Concentration of blood biomarkers predictive of drug efficacy at 6 months and 1 year | baseline, 6 months and 1 year
  Changes in the levels of neuroinflammation indicators, thormbotic inflammation indicators and novel blood-based biomarkers [e.g. phosphodiesterase 3A(PDE3A), transgelin 2(TAGLN2), integrin subunit alpha M(ITGAM), protein phosphatase, Mg2+/Mn2+ dependent 1D(PPM1D)] associated with the prognosis of CSVD compared with baseline levels at 6 months and 1 year.
Changes in white matter integrity at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using Diffusion Tensor Imaging (DTI) with fiber tractography to evaluate the structural integrity of white matter fibre tract.
Changes in functional connectivity networks at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using resting-state functional MRI (rs-fMRI) to measure the temporal correlation and connectivity between brain regions within a specific network.
Changes in neurovascular coupling (imaging biomarker) at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed by combining Arterial Spin Labeling (ASL) and Blood-Oxygen-Level-Dependent (BOLD) fMRI to measure the hemodynamic response following neural activity in specific regions.
Changes in glymphatic function at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using two complementary methods: the Diffusion Tensor Image Analysis Along the Perivascular Space (DTI-ALPS) index, which serves as an imaging proxy for glymphatic system activity, and the quantification of Basal Ganglia Enlarged Perivascular Spaces (BG-EPVS) volume from high-resolution 3D T2-weighted images.
Changes in brain tissue free water at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using multi-compartment Diffusion Tensor Imaging (DTI) models to quantify the fraction of extracellular free water, considered a marker for neuroinflammation and edema.
Changes in heart rate variability (HRV) at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed via analysis of Electrocardiogram (ECG) recordings to evaluate the balance of the autonomic nervous system.
Changes in orthostatic blood pressure at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed via orthostatic testing to measure the cardiovascular system's response to postural changes.
Changes in cerebral autoregulation at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using Transcranial Doppler (TCD) ultrasonography to measure the brain's ability to maintain stable cerebral blood flow despite changes in blood pressure.
Changes in cerebrovascular reactivity at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using Transcranial Doppler (TCD) ultrasonography to measure the dilatory capacity of cerebral blood vessels in response to a vasodilatory stimulus (e.g., CO₂).
Changes in neurovascular coupling (cerebral hemodynamics parameter) at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using task-state Transcranial Doppler (TCD) ultrasonography to measure the relationship between transient neural activity and the subsequent cerebral blood flow response.
Changes in electroencephalography (EEG) oscillatory dispersion at 6 months and 1 year | baseline, 6 months and 1 year
  Assessment of neuroelectrical signals by quantifying the dispersion and variability of oscillatory activity within different EEG frequency bands (e.g., Delta, Theta, Alpha, Beta).
Changes in rey auditory verbal learning test (RAVLT) score at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using the Rey Auditory Verbal Learning Test (RAVLT) to measure memory and learning ability. Performance is scored by the number of words correctly recalled, with scores for a single trial ranging from a minimum of 0 to a maximum of 15. A higher score indicates better performance.
Changes in color trails test (CTT) score at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using the Color Trails Test (CTT) to measure sustained attention and processing speed. Performance is scored by the time required to complete the task. While the theoretical minimum is greater than 0 seconds, the test is typically discontinued if not completed within a maximum cutoff time of 240 seconds. A lower score (faster time) indicates better performance.
Changes in Stroop color and word test (SCWT) score at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using the Stroop Color and Word Test (SCWT) to measure executive function. Performance is scored by the time to completion and the number of errors. The minimum score is 0 seconds and 0 errors. There is no theoretical maximum time, but the maximum number of errors is limited by the total number of items on the test card (e.g., 100 errors on a 100-item card). Lower times and fewer errors indicate better performance.
Changes in verbal fluency test (VFT) score at 6 months and 1 year | baseline, 6 months and 1 year
  Assessed using the Verbal Fluency Test (VFT) to measure language production and executive control. Performance is scored by the total number of correct words generated in a set time. The minimum score is 0, but there is no defined maximum score. A higher score indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, Principal Investigator — Beiling Tiantan Hospital, Capital Medical University

IPD SHARING:
Plan to Share IPD: No